CLINICAL TRIAL: NCT04636762
Title: A Multi-center, Single Arm , Phase II Study of Atezolizumab Combined With Concurrent Chemoradiotherapy and Maintenance Therapy With Atezolizumab in Untreated Participants With Extensive-stage Small Cell Lung Cancer
Brief Title: A Study of Concurrent Chemoradiation With Atezolizumab in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, xianling liu, director of the oncology department of the Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLC-LXL001
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Extensive-stage small cell lung cancer; PD-L1; Atezolizumab; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: To assess safety and tolerability of Atezolizumab Combined with Concurrent Chemoradiotherapy and maintenance therapy with Atezolizumab in untreated participants with extensive-disease small cell lung cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (etoposide, cisplatin, carboplatin, radiation, Atezolizumab) (Experimental): Participants receive EC/EP chemotherapy combined with Atezolizumab（ PD-L1 inhibitor）for 2 cycles, and the efficacy is evaluated 2 weeks after the treatment. If the efficacy evaluation is SD/PR/CR, concurrent chemoradiotherapy with EC/EP(2 cycles) + Atezolizumab） will be initiated. After concurrent chemoradiotherapy+ Atezolizumab, Atezolizumab was maintained until PD or intolerance or for at most 2 years. Participants with brain metastases will receive radiotherapy forbrain metastases during the first 2 cycles of chemotherapy.
  Interventions: Procedure: Radiation Therapy

INTERVENTIONS:
Procedure: Radiation Therapy — Thoracic Radiation Dose: 3Gy, QD, total dose: 30-45Gy; Particpants with brain metastases：metastatic lesions≤3:whole brain radiotherapy with local simultaneous PGTV:50Gy/10F；metastatic lesions>3:whole brain radiotherapy PTV:30Gy/10F.

SUMMARY:
Etoposide-cisplatin/ -carboplatin in combination with PD-L1 inhibitor for 4 cycles followed by maintenance therapy with PD-L1 inhibitor is currently the world-wide first-line treatment for extensive-stage small cell lung cancer. When 4 cycles of EC/EP chemotherapy combined with PD-L1 inhibitor are effective, guidelines recommend additional thoracic radiotherapy.

In our study, the investigators bring radiotherapy forward, which means that after 2 cycles of EC/EP chemotherapy plus Atezolizumab, participants with response（PR/CR/SD）will receive concurrent radiotherapy and 2 cycles of EC/EP chemotherapy plus Atezolizumab, then maintenance therapy with Atezolizumab （Q3W）.

The purpose of this study is to explore the safety and efficacy of Atezolizumab combined with concurrent chemoradiotherapy in untreated participants with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
participants receive EC/EP chemotherapy combined with Atezolizumab for 2 cycles, and the efficacy will be evaluated. If the efficacy evaluation is SD/PR/CR, concurrent chemoradiotherapy comined with EC/EP(2 cycles) +Atezolizumab will be initiated. After concurrent chemoradiotherapy +Atezolizumab, Atezolizumab was maintained until PD or intolerance or for at most 2 years.

participants with brain metastases will receive radiotherapy for brain metastases during the first 2 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1.Histologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system) 2.Must sign a written informed consent form prior to any study specific procedures 3. No prior treatment for ES-SCLC 4.Measurable disease, as defined by RECIST v1.1 5.Can tolerate radiotherapy, no contraindication of radiotherapy 6.Weight≥40kg 7.Life expectancy>12 weeks 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1. 9.Systemic immunosuppressive doses of corticosteroids (prednisone>10 mg/d or equivalent) was discontinued at least 2 weeks before registration for protocol therapy.

10. Be willing to provide 20 tissue sections(4-6 micron thickness) from a newly obtained core or excisional biopsy of a tumor lesion, for biomarker exploration; newly-obtained is defined as a specimen obtained within 3 months before initiation of treatment on day 1; newly-obtained samples must be core needle biopsy, excision, or incision 11.Must have adequate organ function defined by the following laboratory results:

1. Absolute neutrophil count (ANC) ≥ 1.5×109/L, Platelets≥ 100×109/L, Hemoglobin≥90g/L
2. Serum creatinine ≤ 1.5 upper limit of normal (ULN) OR calculated creatinine clearance≥60 mL/min(using Cock-Gault formula)
3. Total bilirubin ≤1.5 ULN or for total bilirubin level ≥1.5 ULN, direct bilirubin is within normal limits; AST (SGOT) and ALT (SGPT)≤2.5 ULN.
4. The thyroid-stimulating hormone (TSH) is within normal range. Note: If the Baseline TSH is not within the normal range, and T3 and T4 are within the normal range, the subject may still meet the inclusion criteria.
5. International normalized ratio(INR) or prothrombin time(PT), activated partial thromboplastin time (APTT)≤1.5 ULN, exception: In subjects receiving anticoagulant therapy, as long as PT or APTT is within the recommended use of anticoagulants
6. Baseline ECG showed no prolonged PR interval or atrioventricular block. 12.Women of child-bearing potential should agree that contraception (such as intrauterine devices(LUD), birth control pills or condoms) must be used during the course of the study through 6 months after the last dose of study medication, and women of childbearing potential should have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication and must be a non-lactation participant; the male participants agree to use contraception during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

1. Hypersensitivity to Atezolizumab
2. Carcinomatous meningitis.
3. History of active Bacillus tuberculosis (TB)
4. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
5. HIV positive or with Acquired Immune Deficiency Syndrome
6. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy
7. History of, or any evidence of active, non-infectious pneumonitis
8. Immunosuppressive drug was used 2 weeks prior to the first study drug treatment, excluding topical glucocorticoid, systematic glucocorticoid not exceeding 10 mg/d of prednisone or equivalent dose of other glucocorticoid
9. Received a live vaccine within 30 days of planned start of study therapy
10. Received a prior anti-cancer monoclonal antibody (mAb) within 3 months prior to study day 1
11. Has taken Chinese herbal medicine for anti-cancer purpose in the past 2 weeks
12. Known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (HCV) (e.g., HCV ribonucleic acid [RNA] [qualitative] is detected)
13. Active infection requiring systemic therapy
14. Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
15. Bleeding tendency, such as active peptic ulcer, or treated with anticoagulants or vitamin K antagonists, such as Warfarin, Heparin, or their analogues
16. Any severe and/or uncontrolled disease, such as: (1) unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months prior to randomization, severe uncontrolled arrhythmia; poor blood pressure control (SBP>140 mmHg, DBP>90 mmHg) ; (2)active or uncontrolled severe infection; (3)liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis; (4) poor control of diabetes (FBG>10mmol/l) ; (5) urine routine suggested urinary protein ≥ + + and 24-hour urinary protein quantitation >1.0 g; (6) history of psychotropic substance abuse and could not be cured or had mental disorder
17. Prisoner who is imprisoned or forcibly detained for reasons other than mental or physical (e.g. infectious) disease
18. Can not tolerate venipuncture
19. Pregnant or lactating women
20. Other conditions that researchers consider unsuitable for participation -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events and the grade of adverse events as assessed by CTCAE v4.0. | 0-36month

SECONDARY OUTCOMES:
Duration of Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1 | 0-120 months
  PFS is defined as the period from the start of receiving the first EC/EP chemotherapy plus PD-L1 inhibitor to disease progression.PFS is assessed by the Investigator Using RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan cancer hospital, Changsha, Hunan
  - the second Xiangya hospital, Changsha, Hunan

REFERENCES:
- [Derived] Liu C, Zeng L, Deng C, Jiang W, Wang Y, Zhou Y, Liu L, Wang S, Zhou C, Qiu Z, Zeng F, Wu F, Weng J, Liu X, Yang N, Ma F. Hypofractionated radiotherapy with immunochemotherapy for extensive-stage small-cell lung cancer. Front Immunol. 2023 Jun 7;14:1175960. doi: 10.3389/fimmu.2023.1175960. eCollection 2023. PMID 37350968